CLINICAL TRIAL: NCT07249723
Title: Comparison of the Effectiveness of Two Active Distraction Methods in Reducing Pain, Fear, and Anxiety in Children Undergoing Venous Blood Sampling
Brief Title: Comparison of the Effectiveness of Two Active Distraction Techniques During Venipuncture in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sinem Yalnızoglu Caka, Assoc. Prof., Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18.11.2025; 2209 (Other Grant/Funding Number: TÜBİTAK)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Nursing Care; Pain Management; Anxiety; Children
Keywords: Acute pain; Distraction; Bubble blowing; Positive reinforcement; Acute pain; Distraction; Bubble blowing; Positive reinforcement
MeSH Terms: conditions — Agnosia; Anxiety Disorders; Acute Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (third party blinding- Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bubble Blowing Group (Experimental): Before the procedure, each child was given a bubble toy and instructed to blow bubbles throughout the procedure. The procedure duration was recorded with a stopwatch. Post-procedural pain and anxiety were assessed using standardized scales. A single-use bubble toy was used for each child.
  Interventions: Other: Bubble Blowing Group
- Positive Reinforcement Group (Experimental): Before the procedure, the researcher established communication with the child, and a short cognitive activity chosen by the child (e.g., counting numbers, word game) was implemented throughout the procedure. The parent provided physical and verbal support to the child. After the procedure, the child received verbal positive reinforcement.
  Interventions: Other: Positive Reinforcement Group
- Standard Procedure Blood Sampling Group (No Intervention): Children in the control group underwent the standard blood sampling procedure in accordance with routine clinical practice. Outcome measurements were conducted after the procedure. Once data collection was completed, children in this group also received verbal feedback. All measurements were performed immediately before and after venipuncture. A single-needle insertion technique was used, and all blood draws were performed by the same pediatric nurse, who was permanently assigned to the unit, to ensure procedural standardization.

INTERVENTIONS:
Other: Bubble Blowing Group — In the Bubble Blowing Group, children were given a bubble toy during the procedure and asked to blow bubbles. This method, which requires active motor participation, was used to divert the children's attention away from the stress of the procedure.
  Arms: Bubble Blowing Group
Other: Positive Reinforcement Group — In the Positive Reinforcement Group, children performed a non-material cognitive activity of their choice during the procedure (such as counting, reciting a short poem/song, or a word game). At the end of the procedure, verbal positive reinforcement was provided (e.g., "Well done," "You were very brave").
  Arms: Positive Reinforcement Group

SUMMARY:
This study was conducted to compare the effects of two active distraction methods-bubble blowing and a material-free cognitive distraction/positive reinforcement technique-applied during venous blood sampling on pain, fear, and anxiety levels in children aged 7-12 years.

DETAILED DESCRIPTION:
Distraction is an effective non-pharmacological nursing intervention used to reduce pain, fear, and anxiety in children during invasive procedures. This approach aims to decrease the child's emotional distress by diverting attention away from the perceived threat.

In particular, among children aged 7-12 years, procedure-related fear and avoidance behaviors may increase due to the impact of previous medical experiences; therefore, there is a need for comparative evaluation of effective distraction strategies tailored to this age group. While sensory-kinesthetic methods such as bubble blowing promote active participation, material-free cognitive techniques can be implemented in any setting and offer easily accessible options. However, studies directly comparing these methods remain limited.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 7 and 12 years,
* Literate (able to read and write),
* Having no diagnosed visual, hearing, intellectual, or neurological disorder,
* With no history of analgesic, sedative, or narcotic use within 24 hours prior to admission,
* Children who, together with their parent, volunteered to participate.

Exclusion Criteria:

* Children who do not meet the inclusion criteria,
* Children or parents who wish to withdraw from the study at any stage,
* Children from whom a blood sample could not be obtained with a single venipuncture attempt.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale (WB-FACES) | A total of 2 evaluations will be made: before the procedure starts, the post-test immediately after the end of the procedure.
  Developed by Wong and Baker (1988), this scale assesses pain intensity in children aged 3-18 years based on facial expressions, using a 0-5 scoring system. Pain intensity was assessed using the Wong-Baker FACES Pain Rating Scale (0-10; higher scores indicate worse pain).
Children's Fear and Anxiety Scale (CFS) | A total of 2 evaluations will be made: before the procedure starts, the post-test immediately after the end of the procedure.
  Developed by McMurtry et al. (2011) and adapted into Turkish by Gerçeker et al. (2018), this scale evaluates fear and anxiety during the procedure on a 0-4 rating scale. 0-10; higher scores indicate greater fear and anxiety.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | A total of 2 evaluations will be made: before the procedure starts, the post-test immediately after the end of the procedure.
  The VAS is a valid and reliable scale that measures pain intensity on a 0-10 cm linear line (Wewers & Lowe, 1990). All scales were administered before and after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Czech O, Wrzeciono A, Rutkowska A, Guzik A, Kiper P, Rutkowski S. Virtual Reality Interventions for Needle-Related Procedural Pain, Fear and Anxiety-A Systematic Review and Meta-Analysis. J Clin Med. 2021 Jul 23;10(15):3248. doi: 10.3390/jcm10153248. PMID 34362032
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Yu Z, Zhou Y, Xu X, Lin L, Le Q, Gu Y. Pharmacological and non-pharmacological interventions in management of peripheral venipuncture-related pain: a randomized clinical trial. BMC Pediatr. 2023 Feb 3;23(1):58. doi: 10.1186/s12887-023-03855-z. PMID 36737707
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] Lawson SL, Hogg MM, Moore CG, Anderson WE, Osipoff PS, Runyon MS, Reynolds SL. Pediatric Pain Assessment in the Emergency Department: Patient and Caregiver Agreement Using the Wong-Baker FACES and the Faces Pain Scale-Revised. Pediatr Emerg Care. 2021 Dec 1;37(12):e950-e954. doi: 10.1097/PEC.0000000000001837. PMID 31335787
- [Background] Inan G, Inal S. The Impact of 3 Different Distraction Techniques on the Pain and Anxiety Levels of Children During Venipuncture: A Clinical Trial. Clin J Pain. 2019 Feb;35(2):140-147. doi: 10.1097/AJP.0000000000000666. PMID 30362982
- [Background] Gerçeker, G.Ö., Ayar, D., Özdemir, E. Z., & Bektaş, M. (2018). Gaining of Children's state anxiety and Children's fear scale to Turkish language. E- Journal of Dokuz Eylul University Nursing Faculty, 11(1), 9-13. https://dergipark.org.tr/tr/pub/deuhfed/issue/46786/586670
- [Background] Erdogan B, Aytekin Ozdemir A. The Effect of Three Different Methods on Venipuncture Pain and Anxiety in Children: Distraction Cards, Virtual Reality, and Buzzy(R) (Randomized Controlled Trial). J Pediatr Nurs. 2021 May-Jun;58:e54-e62. doi: 10.1016/j.pedn.2021.01.001. Epub 2021 Jan 21. PMID 33485746
- [Background] Addab S, Hamdy R, Thorstad K, Le May S, Tsimicalis A. Use of virtual reality in managing paediatric procedural pain and anxiety: An integrative literature review. J Clin Nurs. 2022 Nov;31(21-22):3032-3059. doi: 10.1111/jocn.16217. Epub 2022 Jan 23. PMID 35068011